CLINICAL TRIAL: NCT05900323
Title: Effect of Implementing Enteral Nutrition Guidelines on Critical Care Nurses' Practice and Patients' Outcomes
Brief Title: Enteral Nutrition Guidelines and Patients' Outcomes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, sara Elsayed Ali Hegazy, Assistant Lecturer, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Enteral Nutrition
Record Dates: First submitted 2023-05-29; First posted 2023-06-12 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Enteral Nutrition
Keywords: Enteral nutrition guidelines; Critical care nurses' practice; Patients' outcomes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enteral Nutrition Guidelines Group (Experimental): It will include 34 patients who will receive enteral nutrition guidelines.
  Interventions: Combination Product: enteral nutrition guidelines
- Routine Enteral Nutrition Unit Care Group (No Intervention): It will include 34 patients who will receive routine enteral nutrition unit care.

INTERVENTIONS:
Combination Product: enteral nutrition guidelines — The nurses will be educated about the enteral nutrition guidelines. Then they will apply these guidelines on the participants during enteral nutrition procedure. After conducting the guidelines, the researcher will assess the effect of the guidelines on patients' outcomes.
  Other Names: prokinetic agent
  Arms: Enteral Nutrition Guidelines Group

SUMMARY:
Critically ill patients often exhibit a hypermetabolic state and increased energy requirements due to their critical illnesses. Those patients cannot meet their nutritional requirements through oral feeding. Therefore, the initiation of enteral nutrition (EN) is an essential intervention to fulfill the body's dietary and physiological requirements. Despite advancements in the techniques and equipment used for EN, inadequate nutritional intake is a significant issue for CIPs. It requires special attention to prevent muscle wasting and overfeeding. Critical care nurses have a key role in applying the proper nutritional care for CIPs. They are responsible for inserting and maintaining the feeding tube, delivering the feeds, and avoiding complications associated with EN.

DETAILED DESCRIPTION:
Enteral nutrition is a proactive therapeutic strategy that can be provided by nasogastric or nasoduodenal tubes, gastrostomy, and jejunostomy. It is indicated for the patient who has the digestive capability but is unable to consume enough feeding by mouth. Patients with profound anorexia or severe stress that greatly increases their nutritional needs also require EN. On the other hand, EN is contraindicated for patients with refractory diarrhea, vomiting, bowel obstruction, and when the gastrointestinal tract is not intact.

Despite advancements in the techniques and equipment used for EN, inadequate nutritional intake is a significant issue for CIPs. It requires special attention to prevent muscle wasting and overfeeding. Underfeeding has detrimental effects on patients' clinical outcomes such as delayed wound healing, increased infectious complications, prolonged mechanical ventilation and length of stay in the ICU, and higher mortality rates. Adequate patient nutrition depends on specific interventions or protocols used for planning, initiation, and detection of its complications. Therefore, various nutritional support guidelines are being continuously developed and enriched to help clinical workers improve their nutritional care practice and patients' outcomes.

While the process of administering EN may appear less complex compared with parenteral nutrition, serious complications, and death can result due to potential adverse events occurring throughout the process of ordering, administering, and monitoring EN. These events include reports of metabolic abnormalities, bronchopulmonary aspiration, feeding intolerance, and drug-nutrient interactions.

Because of the significant effects of nursing care on all aspects of EN delivery and management, accurate feeding procedure and avoidance of its associated complications should be considered as a crucial component of nurses' practice. An extensive review of the literature revealed that the patient's clinical outcomes were not evaluated in most studies in Egypt; however, CIPs have a high risk of developing malnutrition or feeding intolerance which is associated with worse clinical outcomes. This inspired us to carry out this study to cover this area.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥ 18 years old.
* Hemodynamically stable patients.
* Patients who are unable to maintain volitional oral intake within 24 hours of admission.

Exclusion Criteria:

* Signs of feeding intolerance (nausea, vomiting, diarrhea, or high gastric residual volume).
* Contraindications to EN such as active bleeding, bowel obstruction, bowel ischemia, or paralytic ileus.
* Signs of clinical shock (low blood pressure, rapid breathing, rapid weak pulse, and decreased urine output).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-01-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Signs of feeding intolerance assessment | Signs of feeding intolerance will be assessed for seven days.
  Absence of vomiting, diarrhea, constipation, abdominal distention, and Normal gastric residual volume.

CONTACTS AND LOCATIONS:
Overall Officials: Sara EA Hegazy, Principal Investigator — Faculty of Nursing, Mansoura University